CLINICAL TRIAL: NCT03579264
Title: Experience and Health Impact of University Students Accessing a Digital Nutrition, Fitness and Mindfulness Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Revive Wellness Inc. (Unknown); Canadian Foundation for Dietetic Research (CFDR) (Other); Mitacs (Industry)
Responsible Party: Principal Investigator, Carla Prado, Associate Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00079680
Record Dates: First submitted 2018-06-13; First posted 2018-07-06 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Stress; Health Behavior; Nutrition; Physical Activity
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Arm (No Intervention): No use of My Viva Plan.
- Intervention Arm (Experimental): Use of My Viva Plan.
  Interventions: Behavioral: My Viva Plan

INTERVENTIONS:
Behavioral: My Viva Plan — Use of the online platform, My Viva Plan, to support health and wellness.
  Arms: Intervention Arm

SUMMARY:
Dietary choices, quality of life and stress will be evaluated in a sample of 100 undergraduate students who are in their first year of university. Students will be randomized into the following two groups; intervention arm (students who will use a preventative self-care program for 12 weeks) vs. control arm (students who will not use a preventative self-care program for 12 weeks).

DETAILED DESCRIPTION:
When individuals look after their own health using online applications they can expect similar or even better health outcomes compared to those obtained by using conventional methods. These kind of tools are popular among University students. Due to the many changes and challenges that students face in the first year of University, this sector of our population is at higher risk of presenting nutritional problems, anxiety, depression and suicidal thoughts.

Recently, a Canadian online application called My Viva Plan® became available. This program is based on preventive self-care and it includes three key pillars of health: nutrition, fitness, and mindfulness. Changes in dietary choices, quality of life and stress will be evaluated in a sample of 100 undergraduate students who are in their first year of university. Students will be randomized into the following two groups; students who will use the program vs. students who will not use the program. Questionnaires regarding physical activity, mindfulness and mental well-being will be evaluated at baseline, week 6 and week 12. Body composition characteristics using bioelectrical impedance analysis will be collected at the start and end of the study (baseline and week 12).

The objective is to determine if the use of an online application based on preventive self-care will result in better food choices, better quality of life, and reduced stress in first year university students.

ELIGIBILITY:
Inclusion Criteria:

* First-year undergraduate university students attending the University of Alberta's North Campus
* Students who are able to complete study assessments in their first year of university
* 17-30 years of age

Exclusion Criteria:

* Students with self-reported eating disorders
* Students with self-reported untreated depression, anxiety or other mood disorders
* Students who do not own a device to access the internet (i.e. tablet, computer, laptop, smart phone)
* Students who are not able to communicate in English
* Pregnant or lactating women
* Individuals with pace-makers or electronic implantable devices

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 97 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Stress | Baseline, week 12
  To assess the change in self reported stress from baseline to week 12 using the Stress Indicators Questionnaire by the International Counselling Team.

SECONDARY OUTCOMES:
Change in Dietary Choices | Baseline, week 12
  To assess the change in dietary choices from baseline to week 12 using three-day food records collected at baseline and week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Prado, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mota JF, Lopes LCC, Trottier CF, Johnson ST, Lieffers J, Prado CM. A Randomized Controlled Trial of the Effects of a Web-Based Intervention on Perceived Stress and Diet Quality Among First-Year University Students. Telemed Rep. 2023 Oct 26;4(1):327-335. doi: 10.1089/tmr.2023.0041. eCollection 2023. PMID 37908625
- [Derived] Lieffers JRL, Quintanilha M, Trottier CF, Johnson ST, Mota JF, Prado CM. Experiences with and Perception of a Web-Based Mindfulness, Nutrition, and Fitness Platform Reported by First-Year University Students: A Qualitative Study. J Acad Nutr Diet. 2021 Dec;121(12):2409-2418.e3. doi: 10.1016/j.jand.2021.04.019. Epub 2021 Jun 10. PMID 34119458
- [Derived] Trottier CF, Lieffers JRL, Johnson ST, Mota JF, Gill RK, Prado CM. The Impact of a Web-Based Mindfulness, Nutrition, and Physical Activity Platform on the Health Status of First-Year University Students: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Mar 10;10(3):e24534. doi: 10.2196/24534. PMID 33688844